CLINICAL TRIAL: NCT03296293
Title: Doctor of Department of Emergency and Critical Care Medicine, Zhoupu Hospital Affiliated With Shanghai University of Medicine and Health Sciences, Shanghai 201318, PR China
Brief Title: Effects of Positive End-expiratory Pressure on Intracranial Pressure in Patients With Severe Traumatic Brain Injury
Acronym: PEEP，ICP，CVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hongpeng Li (Other)
Responsible Party: Sponsor-Investigator, Hongpeng Li, medicine master, Zhoupu Hospital, Pudong New Area, Shanghai, China
Organization: Zhoupu Hospital, Pudong New Area, Shanghai, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZhoupuH
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Brain Injury; Mechanical Ventilation Complication
Keywords: Positive end-expiratory pressure(PEEP); intracranial pressure(ICP); central venous pressure(CVP); intracranial central venous pressure difference(IVPD)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I:IVPD≤3mmHg (Other): Effect of PEEP at 5cmH2O on ICP in Group I:IVPD≤3mmHg Effect of PEEP at 10cmH2O on ICP in Group I:IVPD≤3mmHg Effect of PEEP at 15cmH2O on ICP in Group I:IVPD≤3mmHg
  Interventions: Other: PEEP at 5cmH2O; Other: PEEP at 10cmH2O; Other: PEEP at 15cmH2O
- Group II:3mmHg<IVPD≤6mmHg (Other): Effect of PEEP at 5cmH2O on ICP in Group II:3mmHg<IVPD≤6mmHg Effect of PEEP at 10cmH2O on ICP in Group II:3mmHg<IVPD≤6mmHg Effect of PEEP at 15cmH2O on ICP in Group II:3mmHg<IVPD≤6mmHg
  Interventions: Other: PEEP at 5cmH2O; Other: PEEP at 10cmH2O; Other: PEEP at 15cmH2O
- Group III:IVPD>6mmHg (Other): Effect of PEEP at 5cmH2O on ICP in Group III:IVPD>6mmHg Effect of PEEP at 10cmH2O on ICP in Group III:IVPD>6mmHg Effect of PEEP at 15cmH2O on ICP in Group III:IVPD>6mmHg
  Interventions: Other: PEEP at 5cmH2O; Other: PEEP at 10cmH2O; Other: PEEP at 15cmH2O

INTERVENTIONS:
Other: PEEP at 5cmH2O — Effect of PEEP at 5cmH2O on ICP
Other: PEEP at 10cmH2O — Effect of PEEP at 10cmH2O on ICP
Other: PEEP at 15cmH2O — Effect of PEEP at 15cmH2O on ICP

SUMMARY:
The impact of PEEP on ICP was dependent on the difference between elevated CVP levels and baseline ICP levels. ICP would increase once elevated CVP through PEEP adjustment exceeds the baseline ICP.

DETAILED DESCRIPTION:
all patients were exposed to incremental PEEP levels of 0, 5, 10, and 15cmH2O with 100% of FiO2. The measurements were done bedside on stabilized hemodynamics and intracranial pressure. The measurement was discontinued if the following situation presented and remedies were applied accordingly: (1) CPP < 60 mmHg (norepinephrine at 0.3~1.0μg/kg.min was used); (2) ICP > 25 mmHg (PEEP was restored to 0); (3) increase of pressure plateau > 35 cmH2O (tidal volume was decreased and PetCO2 was maintained at 30~35mmHg); (4) SpO2 < 90% (PEEP was restored to 0); and (5) suspicion of pneumothorax (PEEP was restored to 0 and chest radiography was performed). An equilibration period (at least 90 seconds) was entailed to ensure a normalized baseline PetCO2 through modulating tidal volume and respiratory rate.

ICP, CVP, Pj, and MAP were measured twice or more at each level of PEEP for consecutively five days after admission. CPP was calculated according to the following equation: CPP=MAP-ICP. The difference between baseline ICP and CVP was categorized into the following three groups according to the previous findings: Group I,IVPD ≤ 3mmHg, Group II, 3 < IVPD ≤ 6 mmHg, Group III, IVPD > 6 mmHg. Relationships between PEEP and ICP, CVP and MAP, CVP and Pj were analyzed in each group respectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with sTBI (GCS≤8) and applied with MV were initially included.

Exclusion Criteria:

* Brain death
* Younger than 18 or older than 80 years
* Pregnancy
* Hemodynamic instability：for example heart rate >120 bpm or CPP <60 mmHg
* Bulbous lung or pneumothorax
* Myocardial infarction
* Refusal of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Effects of positive end-expiratory pressure on intracranial pressure in patients with severe traumatic brain injury | up to 12 months
  The impact of PEEP on ICP was dependent on the difference between elevated CVP levels and baseline ICP levels. ICP would increase once elevated CVP through PEEP adjustment exceeds the baseline ICP.

CONTACTS AND LOCATIONS:
Overall Officials: Hongpeng Li, master, Principal Investigator — Department of Emergency and Critical Care Medicine, Zhoupu Hospital affiliated with Shanghai University of Medicine and Health Sciences, Shanghai 201318, PR China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nemer SN, Caldeira JB, Santos RG, Guimaraes BL, Garcia JM, Prado D, Silva RT, Azeredo LM, Faria ER, Souza PC. Effects of positive end-expiratory pressure on brain tissue oxygen pressure of severe traumatic brain injury patients with acute respiratory distress syndrome: A pilot study. J Crit Care. 2015 Dec;30(6):1263-6. doi: 10.1016/j.jcrc.2015.07.019. Epub 2015 Jul 26. PMID 26307004
- [Result] Muench E, Bauhuf C, Roth H, Horn P, Phillips M, Marquetant N, Quintel M, Vajkoczy P. Effects of positive end-expiratory pressure on regional cerebral blood flow, intracranial pressure, and brain tissue oxygenation. Crit Care Med. 2005 Oct;33(10):2367-72. doi: 10.1097/01.ccm.0000181732.37319.df. PMID 16215394
- [Result] Boone MD, Jinadasa SP, Mueller A, Shaefi S, Kasper EM, Hanafy KA, O'Gara BP, Talmor DS. The Effect of Positive End-Expiratory Pressure on Intracranial Pressure and Cerebral Hemodynamics. Neurocrit Care. 2017 Apr;26(2):174-181. doi: 10.1007/s12028-016-0328-9. PMID 27848125
- [Result] Ropper AH, O'Rourke D, Kennedy SK. Head position, intracranial pressure, and compliance. Neurology. 1982 Nov;32(11):1288-91. doi: 10.1212/wnl.32.11.1288. PMID 6890165
- [Result] Shojaee M, Sabzghabaei A, Alimohammadi H, Derakhshanfar H, Amini A, Esmailzadeh B. Effect of Positive End-Expiratory Pressure on Central Venous Pressure in Patients under Mechanical Ventilation. Emerg (Tehran). 2017;5(1):e1. Epub 2017 Jan 8. PMID 28286808

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03296293/Prot_SAP_000.pdf